CLINICAL TRIAL: NCT06430697
Title: Prospective Study Evaluating the Hemodynamic Impact of PAracetamol Administration in Patients Hospitalized in the REAnimation Intensive Care Unit
Brief Title: Hemodynamic Impact of the Administration of PAracetamol in Patients Hospitalized in the Intensive Resuscitation Medicine Department [PAREA]
Acronym: PAREA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-AOI-13
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Intensive Care Unit Syndrome
Keywords: Intensive Care Unit; PARACETAMOL; blood pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with paracetamol (Experimental)
  Interventions: Drug: paracetamol administration

INTERVENTIONS:
Drug: paracetamol administration — Patient hospitalized in Intensive Care Unit with a continuous measurement of blood pressure with a catheter and who have an administration of paracetamol by intravenous or per os

SUMMARY:
Paracetamol is commonly used in case of pain or fever. Few previously clinical studies has highlighted an arterial hypotension linked to intravenous administration of paracetamol. Currently, fewer data are available on the link of intravenous administration of paracetamol and effects on arterial tension. The aim of this study is to describe the frequency of occurrence of significative arterial hypotension within one hour following intravenous or per os administration of paracetamol . Other factors who can be associated to occurence of significative arterial hypotension will be also observe (for example age, weight, pain, vasopressor dosage or sedative...)

ELIGIBILITY:
Inclusion Criteria:

Inclusion:

* 18 years of age or older
* Patient with arterial catheter
* Indication of paracetamol's administration by the patient's attending practitioner.
* No opposition to patient or support person participation in the study if the patient is unable to participate

ExclusionCriteria:

* No Social Security Patient
* Pregnant or nursing patient.
* Patient with a legal protection measure
* Hypersensitivity and/or allergy to paracetamol.
* Contraindication to the use of paracetamol.
* Patient opposition to health data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Measure frequency of low blood pressure following paracetamol administration | One hour after administration of paracetamol
  Proportion of patients with clinically significant low blood pressure occurring within one hour of administration of paracetamol IV or per os. Clinically significant low blood pressure is defined as an average blood pressure of less than 60 mmHg and/or a decrease in average blood pressure of more than 15%, and/or need for vascular filling and/or initiation or increase of the dose of noradrenaline

SECONDARY OUTCOMES:
Measure of blood pressure following paracetamol administration according to IGS II score | One hour after administration of paracetamol
  Identify patients' predictors of low blood pressure following paracetamol administration : Patients' will be identified by measuring frequency of patients with low blood pressure following paracetamol administration, according to The IGS II score (Simplified Severity Index II) is a score used to assess the severity of a patient and is one of the scores used in intensive care and SOFA score.
  Components: The IGS II includes several variables, such as age, chronic health conditions, vital signs, and laboratory values. These factors are combined to calculate a numerical score.
  Scoring: The higher the IGS II score, the greater the predicted risk of mortality. The score ranges from 0 to 100, with higher values indicating more severe illness.
identify predictors linked to paracetamol administration route | One hour after administration of paracetamol
  Measure of blood pressure to identify predictors by measuring frequency of patients with low blood pressure following paracetamol administration, according to administration's route
identify predictors linked to paracetamol dosage | One hour after administration of paracetamol
  Measure of blood pressure to identify predictors by measuring frequency of patients with low blood pressure following paracetamol administration, according to dosage
Measure of blood pressure following paracetamol administration according to SOFA score | One hour after administration of paracetamol
  Identify patients' predictors of low blood pressure following paracetamol administration : Patients' will be identified by measuring frequency of patients with low blood pressure following paracetamol administration, according to the SOFA score.
  The sequential organ failure assessment score (SOFA score), previously known as the sepsis-related organ failure assessment score,is used to track a person's status during the stay in an intensive care unit (ICU) to determine the extent of a person's organ function or rate of failure.
  Each system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). The worst physiological variables are collected serially every 24 hours of a patient's ICU admission12. The total SOFA score ranges from 0 (best) to 24 (worst) points. It's a valuable tool for predicting clinical outcomes in critically ill patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE ARCHET, Nice, France